CLINICAL TRIAL: NCT03564353
Title: Investigating Memory in Healthy Subjects Using Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-34 CM
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adults
Keywords: transcranial Direct Current Stimulation (tDCS); memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four groups: (1) tDCS targeting location 1 paired with memory task (2) tDCS targeting location 2 with memory task (3) tDCS targeting location 3 paired with memory task (4) tDCS targeting location 4 paired with memory task
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- memory task with tDCS location 1 (Experimental): memory task paired with tDCS targeting C2 nerve (anode left c2; cathode right C2)
  Interventions: Device: tDCS
- memory task with tDCS location 2 (Experimental): memory task paired with tDCS targeting C2 nerve (anode right c2; cathode left C2)
  Interventions: Device: tDCS
- memory task with tDCS location 3 (Experimental): memory task paired with tDCS targeting C5/6 nerve
  Interventions: Device: tDCS
- memory task with tDCS location 4 (Experimental): memory task paired with tDCS targeting trigeminal nerve dermatomes (left and right temple/jaw)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS

SUMMARY:
The purpose of this study is to investigate whether we can improve associative memory performance in healthy subjects, by applying transcranial Direct Current Stimulation (tDCS) during a verbal paired-associate learning task

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer's disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Transcranial Direct Current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has demonstrated to accelerate learning and improve memory in some studies. To investigate whether it is possible to improve associative memory using tDCS, the performance in a Verbal Paired-Associate memory task of 4 groups targeting different areas will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Native English Speaker

Exclusion Criteria:

* History of severe head injuries, epileptic insults, or heart disease.
* Severe psychiatric disorders and severe untreated medical problems.
* acquainted with the foreign language used in the learning task
* Contraindications for tDCS (pregnant women, implanted devices)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas of Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- C2 Right: memory task paired with tDCS targeting the right Cranial 2 Nerve (C2) using anodal stimulation
  tDCS: tDCS
- C2 Left: memory task paired with tDCS targeting the left Cranial 2 (C2) nerve using anodal stimulation
  tDCS: tDCS
- Trigeminal Nerve: memory task paired with tDCS targeting the Trigeminal Nerve
  tDCS: tDCS
- Cranial 5/6 Nerves: memory task paired with tDCS targeting the fifth cranial nerve (C5)
  tDCS: tDCS
Period: Overall Study
Arm/Group | C2 Right | C2 Left | Trigeminal Nerve | Cranial 5/6 Nerves
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C2 Right | C2 Left | Trigeminal Nerve | Cranial 5/6 Nerves | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (2.64) | 20.6 (2.17) | 22.8 (4.6) | 22.7 (4.54) | 21.75 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 5 | 21
  Male | 5 | 4 | 5 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This was not collected Population: That was not collected
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data was not colelcted Population: Data was not collected
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Beck Depression Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  The Beck Depression Inventory uses the following scale to assess patients: 0 - 13: Minimal depression, 14 - 19: Mild depression, 20 - 28: Moderate depression, 29 - 63: Severe depression Min score: 0; Max Score: 63; The higher the score the more mood
  units on a scale | 4.1 (4.3) | 4.6 (4.43) | 2.6 (3.9) | 4.9 (4.33) | 4.05 (4.21)
Beck Anxiety Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are:
  0-7: minimal anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
  units on a scale | 7 (13.02) | 2.9 (4.5) | 1.6 (1.95) | 2.6 (3.3) | 3.53 (7.18)
Mini Mental State Examination >25 [Count of Participants; unit: Participants] — Measure Description: The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
  Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
  Participants | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Associative Memory Assessed by a Verbal Paired-Associate Test
Description: Participants got the opportunity to learn the list of 75-word pairs across a total of eight alternating study (S) and test (T) periods. Participants came back for a final test session (all 75 words tested) 7 days later and were asked to give the English translations of Swahili words. A score was calaculated based on the percentage of words (English trnaslations) correctly recalled words.
Time Frame: Baseline and 1 week after the tDCS
Measure: Mean (Standard Error); unit: percentage
Arm/Group | C2 Right | C2 Left | Trigeminal Nerve | Cranial 5/6 Nerves
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage | 50.6 (6.88) | 50.78 (6.88) | 32.77 (6.88) | 30.25 (6.88)

ADVERSE EVENTS:
Time Frame: two weeks
Description: TES Adverse events. We use the tDCS Exit questionnaire developed by Brunoni et al. (36) to assess potential side-effect (headache, neck pain, scalp pain, tingling, itching, burning sensation, skin redness, sleepiness, trouble concentrating, mood changes).
Groups:
- Memory Task With tDCS Location 1: memory task paired with tDCS targeting location 1
  tDCS: tDCS
- Memory Task With tDCS Location 2: memory task paired with tDCS targeting location 2
  tDCS: tDCS
- Memory Task With tDCS Location 3: memory task paired with tDCS targeting location 3
  tDCS: tDCS
- Memory Task With tDCS Location 4: memory task paired with tDCS targeting location 4
  tDCS: tDCS
Arm/Group | Memory Task With tDCS Location 1 | Memory Task With tDCS Location 2 | Memory Task With tDCS Location 3 | Memory Task With tDCS Location 4
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03564353/Prot_002.pdf